CLINICAL TRIAL: NCT02792933
Title: Localization of the Epidural Space Using the Loss of Resistance Technique for Labour Analgesia: A Randomized Controlled Trial Comparing Air Versus Saline Solution
Brief Title: Air Versus Saline Solution for the Localization of the Epidural Space in Labour Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: HULP2914
Record Dates: First submitted 2016-05-10; First posted 2016-06-08 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Effects of Anesthesia Spinal and Epidural in Pregnancy
MeSH Terms: interventions — Air; Injections, Epidural; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- air in epidural space (Active Comparator): When the ALOR epidural localization technique will be used, an intermittent pressure with fast movements will be exerted on the plunger of the syringe while the Tuohy needle will be inserted until loss of resistance was felt.
  Interventions: Procedure: air in epidural space
- saline in epidural space (Experimental): When the SLOR technique is used, a continuous pressure will be exerted on the plunger of the Tuohy needle until loss of resistance was felt.
  Interventions: Procedure: saline in epidural space

INTERVENTIONS:
Procedure: air in epidural space — The epidural puncture will be performed in the L3-L4 or L4-L5 interspinous space in a seated position. A local anaesthesia with 2-5 mL of 2% lidocaine will be applied subcutaneously using a 25Gm 25mm needle. The epidural space will be localized using a Perifix® set by inserting the Tuohy needle in the ligamentum flavum or the interspinous space. The obturator will be then withdrawn and the low resistance syringe filled with 3-5mL of air will be connected. After localizing the epidural space, the catheter will be inserted 3-5 cm. An aspiration test will be performed through the catheter in a decline position with a 2 mL syringe, and a 3mL test dose with bupivacaine 0,25% plus epinephrine 1/200.000 will be administered to exclude an intradural or an intravascular position of the catheter.
  Arms: air in epidural space
Procedure: saline in epidural space — The epidural puncture will be performed in the L3-L4 or L4-L5 interspinous space in a seated position. A local anaesthesia with 2-5 mL of 2% lidocaine will be applied subcutaneously using a 25Gm 25mm needle. The epidural space will be localized using a Perifix® set by inserting the Tuohy needle in the ligamentum flavum or the interspinous space. The obturator will be withdrawn and the low resistance syringe filled with 3-5mL of saline solution will be connected. After localizing the epidural space, the catheter will be inserted 3-5 cm. An aspiration test will be performed through the catheter in a decline position with a 2 mL syringe, and a 3mL test dose with bupivacaine 0,25% plus epinephrine 1/200.000 will be administered to exclude an intradural or an intravascular position of the catheter.
  Arms: saline in epidural space

SUMMARY:
Epidural space localization using loss of resistance technique with air (ALOR) is controversial in obstetric analgesia due to a minor efficacy and risk of complications, compared with loss of resistance technique with saline (SLOR). This randomized prospective study will compare the efficacy and incidence of most common complications of both techniques in obstetric analgesia.

DETAILED DESCRIPTION:
A local ethics committee has approved the study. A statistical power calculation was performed and 177 patients per group will be necessary to confirm a 20% difference of efficacy of the block at 30 minutes (α=0,05; β=0,1). Epidural catheter will be inserted and a standardized analgesic protocol will initiate. The efficacy of the block will be assessed after 30 minutes and at delivery. The apparition of adverse effects during puncture and labour will be annotated. The need for repuncture of the block and the repercussion of the technique on the delivery and the fetus will be recorded as well. At 24 hours, investigators will assess the incidence of pain at the site of puncture (PSP) and the level of maternal satisfaction on a 0 to10 numeric scale.

ELIGIBILITY:
Inclusion criteria:

* Parturients asking for epidural analgesia during labour .
* Age between 18 and 45 years.
* Spontaneous or induced.
* Cervical dilatation inferior to 6 cm.
* Written informed consent.

Exclusion criteria:

* Infection in the puncture site.
* Refusal of the patient.
* Coagulopathy.
* Severe hypovolaemia.
* Intracranial hypertension.
* Severe aortic or mitral stenosis.
* Systemic infection.
* Non collaborating patient.
* Incapacity of communicating or lack of comprehension of the study by the parturient
* Prior neurological symptoms or demyelinising lesions.
* Valvular stenosis.
* Severe spinal deviation.
* Patient previously operated of spinal surgery in the site of puncture.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2009-07; Primary Completion 2010-02 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Analgesia obtained 30 minutes after the puncture of the epidural block (variation of pain score) | 30 min

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Antibas PL, do Nascimento Junior P, Braz LG, Vitor Pereira Doles J, Modolo NS, El Dib R. Air versus saline in the loss of resistance technique for identification of the epidural space. Cochrane Database Syst Rev. 2014 Jul 18;2014(7):CD008938. doi: 10.1002/14651858.CD008938.pub2. PMID 25033878